CLINICAL TRIAL: NCT05576545
Title: Develop and Evaluate the Effectiveness of a Self-Care Smartphone Application on the Self-Efficacy, and Resilience Among Newly Diagnosed Breast Cancer Patients Undergoing Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hsin-Tien Hsu, Principal investigator, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KMUHIRB-E(I)-20200041
Record Dates: First submitted 2022-09-26; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Breast Neoplasm; Breast Malignant Tumor; Resilience; Self-efficacy
Keywords: Breast cancer; mobile application; Resilience; self-efficacy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general routine care and the Breast Cancer Self-Care App (Experimental)
  Interventions: Device: The Breast Cancer Self-Care App
- general routine care (No Intervention)

INTERVENTIONS:
Device: The Breast Cancer Self-Care App — The Breast Cancer Self-Care App includes several parts- introduction to breast cancer, types of treatment, side effects care, nutrition, relaxation videos, insurance, medical news and recording side effects, etc. The researcher assisted in installing the App on the patient's mobile phone, entered the personal account, and asked the patient to fill in questionnaires. Patients were given individual health education task in the Breast Cancer Self-Care App every week according to the type of chemotherapy drugs. After four weeks, they filled in questionnaires again.
  Arms: general routine care and the Breast Cancer Self-Care App

SUMMARY:
This study was to develop and evaluate the self-efficacy and resilience of the Breast Cancer Self-Care App in newly diagnosed breast cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
This study was to develop and evaluate the self-efficacy and resilience of the Breast Cancer Self-Care App in newly diagnosed breast cancer patients undergoing chemotherapy. In the first phase of this study, develop a prototype the Breast Cancer Self-Care App by conducting patients interviews. In the second phase, an experimental two-group pretest-posttest quantitative study design to evaluate the self-efficacy and resilience of the Breast Cancer Self-Care App in newly diagnosed breast cancer patients undergoing chemotherapy. The patients were randomized to the experimental and control groups. Patients in the control group received general routine care and patients in the experimental group received general routine care plus the Breast Cancer Self-Care App intervention. Both groups completed a basic demographics, self-efficacy and resilience questionnaires at the pre-test and after four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Consciousness clear, over 20 years old, can communicate in Mandarin and Taiwanese
* Diagnosed Breast Cancer I-III stage
* undergo first chemotherapy
* Have a smartphone
* Receiving treatment: EC/ EC+T/LC/LC+T E: (Epirubicin)、C: (Cyclophosphamide)、L: (Lipo-Dox)、T: (Taxotere)

Exclusion Criteria:

* DSM-V mentally ill
* IOS system smartphone
* over 65 years old

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | 4 weeks
  Use Strategies Used by People to Promote Health (SUPPH) measure self-care self-efficacy. The scale total of 29 items measure self-care self-efficacy. There are 3 sub subscales for each of the following: Stress Reduction (10 items, 5-50scores), Making Decisions (3 items, 3-15scores), Positive Attitude (16 items,16-80 scores). The range of total scores of the scale is 29-145. It shows that self-care self-efficacy increases as total points of the scale increase.

SECONDARY OUTCOMES:
Resilience | 4 weeks
  Use Resilience scale 14 items (RS-14) measure individual resilience. The scale with a total of 14 items measures resilience. The range of total scores of the scale is 14-98. It shows that resilience increases as total points of the scale increase.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aizpurua-Perez I, Perez-Tejada J. Resilience in women with breast cancer: A systematic review. Eur J Oncol Nurs. 2020 Dec;49:101854. doi: 10.1016/j.ejon.2020.101854. Epub 2020 Oct 10. PMID 33120216
- [Background] Ajčević, M., Dea, F. D., Barbieri, G., & Accardo, A. (2019). A mobile app for the self-management of type 1 diabetes as tool for preventing of exercise-associated glycemic imbalances. World Congress on Medical Physics and Biomedical Engineering 475-479. https://doi.org/10.1007/978-981-10-9035-6_88
- [Background] Akin S, Can G, Durna Z, Aydiner A. The quality of life and self-efficacy of Turkish breast cancer patients undergoing chemotherapy. Eur J Oncol Nurs. 2008 Dec;12(5):449-56. doi: 10.1016/j.ejon.2008.07.006. Epub 2008 Oct 7. PMID 18842460
- [Background] Akin S, Kas Guner C. Investigation of the relationship among fatigue, self-efficacy and quality of life during chemotherapy in patients with breast, lung or gastrointestinal cancer. Eur J Cancer Care (Engl). 2019 Jan;28(1):e12898. doi: 10.1111/ecc.12898. Epub 2018 Jul 24. PMID 30039883
- [Background] Aungst TD, Clauson KA, Misra S, Lewis TL, Husain I. How to identify, assess and utilise mobile medical applications in clinical practice. Int J Clin Pract. 2014 Feb;68(2):155-62. doi: 10.1111/ijcp.12375. PMID 24460614
- [Background] Awan A, Esfahani K. Endocrine therapy for breast cancer in the primary care setting. Curr Oncol. 2018 Aug;25(4):285-291. doi: 10.3747/co.25.4139. Epub 2018 Aug 14. PMID 30111969
- [Background] Ayyoubzadeh SM, Shirkhoda M, R Niakan Kalhori S, Mohammadzadeh N, Zakerabasali S. A Smartphone Remote Monitoring App to Follow Up Colorectal Cancer Survivors: Requirement Analysis. JMIR Cancer. 2022 Jan 5;8(1):e18083. doi: 10.2196/18083. PMID 34989685
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Bandura, A. (1982). Self-efficacy mechanism in human agency. American psychologist, 37(2), 122. https://doi.org/10.1037/0003-066X.37.2.122
- [Background] Bandura, A. (1986). The explanatory and predictive scope of self-efficacy theory. Journal of Social and Clinical Psychology, 4(3), 359-373. https://doi.org/10.1521/jscp.1986.4.3.359
- [Background] Bandura, A. (2010). Self-efficacy the corsini encyclopedia of psychology. John Wiley & Sons, 10, 1-3. https://doi.org/10.1002/9780470479216.corpsy0836
- [Background] Bandura, A., Freeman, W., & Lightsey, R. (1999). Self-efficacy: The exercise of control. 15-17. https://doi.org/10.1007/BF02352723
- [Background] Baumel A, Torous J, Edan S, Kane JM. There is a non-evidence-based app for that: A systematic review and mixed methods analysis of depression- and anxiety-related apps that incorporate unrecognized techniques. J Affect Disord. 2020 Aug 1;273:410-421. doi: 10.1016/j.jad.2020.05.011. Epub 2020 May 11. PMID 32560936
- [Background] Britton WB. Can mindfulness be too much of a good thing? The value of a middle way. Curr Opin Psychol. 2019 Aug;28:159-165. doi: 10.1016/j.copsyc.2018.12.011. Epub 2019 Jan 7. PMID 30708288
- [Background] Buneviciene I, Mekary RA, Smith TR, Onnela JP, Bunevicius A. Can mHealth interventions improve quality of life of cancer patients? A systematic review and meta-analysis. Crit Rev Oncol Hematol. 2021 Jan;157:103123. doi: 10.1016/j.critrevonc.2020.103123. Epub 2020 Oct 20. PMID 33190065
- [Background] Cai T, Huang Y, Zhang Y, Lu Z, Huang Q, Yuan C. Mobile health applications for the care of patients with breast cancer: A scoping review. Int J Nurs Sci. 2021 Aug 25;8(4):470-476. doi: 10.1016/j.ijnss.2021.07.003. eCollection 2021 Oct 10. PMID 34631997
- [Background] Callaghan DM. Health-promoting self-care behaviors, self-care self-efficacy, and self-care agency. Nurs Sci Q. 2003 Jul;16(3):247-54. doi: 10.1177/0894318403016003016. PMID 12876883
- [Background] Chen YC, Huang HM, Kao CC, Sun CK, Chiang CY, Sun FK. The Psychological Process of Breast Cancer Patients Receiving Initial Chemotherapy: Rising From the Ashes. Cancer Nurs. 2016 Nov/Dec;39(6):E36-E44. doi: 10.1097/NCC.0000000000000331. PMID 26713500
- [Background] Chen HL, Liu K, You QS. Self-efficacy, cancer-related fatigue, and quality of life in patients with resected lung cancer. Eur J Cancer Care (Engl). 2018 Nov;27(6):e12934. doi: 10.1111/ecc.12934. Epub 2018 Sep 25. PMID 30252973
- [Background] Chirico A, Lucidi F, Merluzzi T, Alivernini F, Laurentiis M, Botti G, Giordano A. A meta-analytic review of the relationship of cancer coping self-efficacy with distress and quality of life. Oncotarget. 2017 May 30;8(22):36800-36811. doi: 10.18632/oncotarget.15758. PMID 28404938
- [Background] Chou YH, Chia-Rong Hsieh V, Chen X, Huang TY, Shieh SH. Unmet supportive care needs of survival patients with breast cancer in different cancer stages and treatment phases. Taiwan J Obstet Gynecol. 2020 Mar;59(2):231-236. doi: 10.1016/j.tjog.2020.01.010. PMID 32127143
- [Background] Civilotti C, Acquadro Maran D, Santagata F, Varetto A, Stanizzo MR. The use of the Distress Thermometer and the Hospital Anxiety and Depression Scale for screening of anxiety and depression in Italian women newly diagnosed with breast cancer. Support Care Cancer. 2020 Oct;28(10):4997-5004. doi: 10.1007/s00520-020-05343-x. Epub 2020 Feb 8. PMID 32036468
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Daly RM, Gianoudis J, Hall T, Mundell NL, Maddison R. Feasibility, Usability, and Enjoyment of a Home-Based Exercise Program Delivered via an Exercise App for Musculoskeletal Health in Community-Dwelling Older Adults: Short-term Prospective Pilot Study. JMIR Mhealth Uhealth. 2021 Jan 13;9(1):e21094. doi: 10.2196/21094. PMID 33439147
- [Background] Deng G. Integrative Medicine Therapies for Pain Management in Cancer Patients. Cancer J. 2019 Sep/Oct;25(5):343-348. doi: 10.1097/PPO.0000000000000399. PMID 31567462
- [Background] Eberle C, Lohnert M, Stichling S. Effectiveness of Disease-Specific mHealth Apps in Patients With Diabetes Mellitus: Scoping Review. JMIR Mhealth Uhealth. 2021 Feb 15;9(2):e23477. doi: 10.2196/23477. PMID 33587045
- [Background] Eller LS, Lev EL, Yuan C, Watkins AV. Describing Self-Care Self-Efficacy: Definition, Measurement, Outcomes, and Implications. Int J Nurs Knowl. 2018 Jan;29(1):38-48. doi: 10.1111/2047-3095.12143. Epub 2016 May 31. PMID 27245100
- [Background] Fanchiang YC, Yen YH, Chen SW. [Using Nursing Digital Technology to Reduce the Rates of Catheter-Associated and Non-Catheter-Associated Urinary Tract Infection]. Hu Li Za Zhi. 2019 Apr;66(2):77-84. doi: 10.6224/JN.201904_66(2).10. Chinese. PMID 30924517
- [Background] Fang SY, Wang YL, Lu WH, Lee KT, Kuo YL, Fetzer SJ. Long-term effectiveness of an E-based survivorship care plan for breast cancer survivors: A quasi-experimental study. Patient Educ Couns. 2020 Mar;103(3):549-555. doi: 10.1016/j.pec.2019.09.012. Epub 2019 Sep 12. PMID 31558323
- [Background] Fini, I. A., Adib-Hajbaghery, M., & Khachian, A. (2011). The effect of health-promotion strategies education on self-care self-efficacy in patients with bone marrow transplantation. Iranian Journal of Critical Care Nursing, 4(3), 42-44. https://doi.org/10.1038/bmt.2008.113
- [Background] Fisusi FA, Akala EO. Drug Combinations in Breast Cancer Therapy. Pharm Nanotechnol. 2019;7(1):3-23. doi: 10.2174/2211738507666190122111224. PMID 30666921
- [Background] Gagnon MP, Ngangue P, Payne-Gagnon J, Desmartis M. m-Health adoption by healthcare professionals: a systematic review. J Am Med Inform Assoc. 2016 Jan;23(1):212-20. doi: 10.1093/jamia/ocv052. Epub 2015 Jun 15. PMID 26078410
- [Background] Garcia-Dia MJ, DiNapoli JM, Garcia-Ona L, Jakubowski R, O'Flaherty D. Concept analysis: resilience. Arch Psychiatr Nurs. 2013 Dec;27(6):264-70. doi: 10.1016/j.apnu.2013.07.003. Epub 2013 Sep 24. PMID 24238005
- [Background] Giuliano AE, Edge SB, Hortobagyi GN. Eighth Edition of the AJCC Cancer Staging Manual: Breast Cancer. Ann Surg Oncol. 2018 Jul;25(7):1783-1785. doi: 10.1245/s10434-018-6486-6. Epub 2018 Apr 18. No abstract available. PMID 29671136
- [Background] Godfrey CM, Harrison MB, Lysaght R, Lamb M, Graham ID, Oakley P. Care of self - care by other - care of other: the meaning of self-care from research, practice, policy and industry perspectives. Int J Evid Based Healthc. 2011 Mar;9(1):3-24. doi: 10.1111/j.1744-1609.2010.00196.x. PMID 21332659
- [Background] Habibullah G, Gul R, Cassum S, Elahi R. Experiences of the Breast Cancer Patients Undergoing Radiotherapy at a Public Hospital Peshawar Pakistan. Asia Pac J Oncol Nurs. 2018 Apr-Jun;5(2):184-194. doi: 10.4103/apjon.apjon_70_17. PMID 29607379
- [Background] Harrison, R., Flood, D., & Duce, D. (2013). Usability of mobile applications: literature review and rationale for a new usability model. Journal of Interaction Science, 1(1), 1-16. https://doi.org/10.1186/2194-0827-1-1
- [Background] Hou IC, Lin HY, Shen SH, Chang KJ, Tai HC, Tsai AJ, Dykes PC. Quality of Life of Women After a First Diagnosis of Breast Cancer Using a Self-Management Support mHealth App in Taiwan: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Mar 4;8(3):e17084. doi: 10.2196/17084. PMID 32130181
- [Background] Inan FS, Gunusen NP, Ustun B. Experiences of Newly Diagnosed Breast Cancer Patients in Turkey. J Transcult Nurs. 2016 May;27(3):262-9. doi: 10.1177/1043659614550488. Epub 2014 Sep 15. PMID 25225235
- [Background] Jongerius C, Russo S, Mazzocco K, Pravettoni G. Research-Tested Mobile Apps for Breast Cancer Care: Systematic Review. JMIR Mhealth Uhealth. 2019 Feb 11;7(2):e10930. doi: 10.2196/10930. PMID 30741644
- [Background] Kewan T, Alomari M, Khazaaleh S, Covut F, Olayan M. Hand-foot Syndrome Secondary to Low-dose Docetaxel in a Breast Cancer Patient. Cureus. 2019 Apr 6;11(4):e4400. doi: 10.7759/cureus.4400. PMID 31245190
- [Background] Konaszewski, K., Kolemba, M., & Niesiobędzka, M. (2021). Resilience, sense of coherence and self-efficacy as predictors of stress coping style among university students. Current Psychology, 40(8), 4052-4062. https://doi.org/10.1007/s12144-019-00363-1
- [Background] Latifi M, Alishan Karami N, Beiraghdar M, Maraki F, Allahbakhshian Farsani L. Impact of Health Information Prescription on Self-care of Women with Breast Cancer. Adv Biomed Res. 2018 Oct 31;7:139. doi: 10.4103/abr.abr_142_18. eCollection 2018. PMID 30505810
- [Background] Lee TY, Hsing SC, Li CC. An Improved Stress-Scale Specifically Designed to Measure Stress of Women with Newly Diagnosed Breast Cancer. Int J Environ Res Public Health. 2021 Feb 27;18(5):2346. doi: 10.3390/ijerph18052346. PMID 33673627
- [Background] Lin PJ, Fang SY, Kuo YL. Development and Usability Testing of a Decision Support App for Women Considering Breast Reconstruction Surgery. J Cancer Educ. 2021 Feb;36(1):160-167. doi: 10.1007/s13187-019-01612-4. PMID 31463810
- [Background] Lozano-Lozano M, Galiano-Castillo N, Martin-Martin L, Pace-Bedetti N, Fernandez-Lao C, Arroyo-Morales M, Cantarero-Villanueva I. Monitoring Energy Balance in Breast Cancer Survivors Using a Mobile App: Reliability Study. JMIR Mhealth Uhealth. 2018 Mar 27;6(3):e67. doi: 10.2196/mhealth.9669. PMID 29588273
- [Background] Meric-Bernstam F, Johnson AM, Dumbrava EEI, Raghav K, Balaji K, Bhatt M, Murthy RK, Rodon J, Piha-Paul SA. Advances in HER2-Targeted Therapy: Novel Agents and Opportunities Beyond Breast and Gastric Cancer. Clin Cancer Res. 2019 Apr 1;25(7):2033-2041. doi: 10.1158/1078-0432.CCR-18-2275. Epub 2018 Nov 15. PMID 30442682
- [Background] Messner, E.-M., Probst, T., O'Rourke, T., Stoyanov, S., & Baumeister, H. (2019). mHealth applications: potentials, limitations, current quality and future directions. In Digital Phenotyping and Mobile Sensing (pp. 235-248). Springer. https://doi.org/10.1007/978-3-030-31620-4_15
- [Background] Moszeik, E. N., von Oertzen, T., & Renner, K.-H. (2020). Effectiveness of a short Yoga Nidra meditation on stress, sleep, and well-being in a large and diverse sample. Current Psychology, 1-15. https://link.springer.com/article/10.1007/s12144-020-01042-2
- [Background] Omran S, Mcmillan S. Symptom Severity, Anxiety, Depression, Self- Efficacy and Quality of Life in Patients with Cancer. Asian Pac J Cancer Prev. 2018 Feb 26;19(2):365-374. doi: 10.22034/APJCP.2018.19.2.365. PMID 29479979
- [Background] Osborn J, Ajakaiye A, Cooksley T, Subbe CP. Do mHealth applications improve clinical outcomes of patients with cancer? A critical appraisal of the peer-reviewed literature. Support Care Cancer. 2020 Mar;28(3):1469-1479. doi: 10.1007/s00520-019-04945-4. Epub 2019 Jul 4. PMID 31273501
- [Background] Pez M, Keller A, Welzel G, Abo-Madyan Y, Ehmann M, Tuschy B, Berlit S, Sutterlin M, Wenz F, Giordano FA, Sperk E. Long-term outcome after intraoperative radiotherapy as a boost in breast cancer. Strahlenther Onkol. 2020 Apr;196(4):349-355. doi: 10.1007/s00066-019-01525-7. Epub 2019 Oct 22. PMID 31641788
- [Background] Riegel B, Jaarsma T, Stromberg A. A middle-range theory of self-care of chronic illness. ANS Adv Nurs Sci. 2012 Jul-Sep;35(3):194-204. doi: 10.1097/ANS.0b013e318261b1ba. PMID 22739426
- [Background] Sheu, H.-B., Lent, R. W., Miller, M. J., Penn, L. T., Cusick, M. E., & Truong, N. N. (2018). Sources of self-efficacy and outcome expectations in science, technology, engineering, and mathematics domains: A meta-analysis. Journal of Vocational Behavior, 109, 118-136. https://doi.org/10.1016/j.jvb.2018.10.003
- [Background] Sisto A, Vicinanza F, Campanozzi LL, Ricci G, Tartaglini D, Tambone V. Towards a Transversal Definition of Psychological Resilience: A Literature Review. Medicina (Kaunas). 2019 Nov 16;55(11):745. doi: 10.3390/medicina55110745. PMID 31744109
- [Background] Sohrabei, S., & Atashi, A. (2021). The impact of mobile health on breast cancer patient's life and treatment: A systematic review. Frontiers in Health Informatics, 10(1), 88. https://doi.org/10.30699/fhi.v10i1.295
- [Background] Tan WS, Beatty L, Koczwara B. Do cancer patients use the term resilience? A systematic review of qualitative studies. Support Care Cancer. 2019 Jan;27(1):43-56. doi: 10.1007/s00520-018-4456-y. Epub 2018 Sep 12. PMID 30209600
- [Background] van Seijen M, Lips EH, Thompson AM, Nik-Zainal S, Futreal A, Hwang ES, Verschuur E, Lane J, Jonkers J, Rea DW, Wesseling J; PRECISION team. Ductal carcinoma in situ: to treat or not to treat, that is the question. Br J Cancer. 2019 Aug;121(4):285-292. doi: 10.1038/s41416-019-0478-6. Epub 2019 Jul 9. PMID 31285590
- [Background] Wagnild GM, Young HM. Development and psychometric evaluation of the Resilience Scale. J Nurs Meas. 1993 Winter;1(2):165-78. PMID 7850498
- [Background] Wang Z, Cheng Y, Li J, Hu X. Effect of integrated medical and nursing intervention model on quality of life and unhealthy emotion of patients with esophageal cancer undergoing radiotherapy. Am J Transl Res. 2021 Apr 15;13(4):3780-3786. eCollection 2021. PMID 34017565
- [Background] Wang Z, Yin G, Jia R. Impacts of self-care education on adverse events and mental health related quality of life in breast cancer patients under chemotherapy. Complement Ther Med. 2019 Apr;43:165-169. doi: 10.1016/j.ctim.2019.01.027. Epub 2019 Feb 1. PMID 30935525
- [Background] Xu, Y. F., Xu, X. F., Song, K., Qiu, C., Zhang, X., & DI LI NU ER-RE, H. (2021). Effects of Extended Care Based on the WeChat Platform on Self-Efficacy and Quality of Life of Postoperative Breast Cancer Patients. Indian Journal of Pharmaceutical Sciences, 23-30. https://doi.org/10.36468/pharmaceutical-sciences.spl.165
- [Background] Zhou K, Li J, Li X. Effects of cyclic adjustment training delivered via a mobile device on psychological resilience, depression, and anxiety in Chinese post-surgical breast cancer patients. Breast Cancer Res Treat. 2019 Nov;178(1):95-103. doi: 10.1007/s10549-019-05368-9. Epub 2019 Jul 24. PMID 31342310
- [Background] Zhu J, Ebert L, Liu X, Wei D, Chan SW. Mobile Breast Cancer e-Support Program for Chinese Women With Breast Cancer Undergoing Chemotherapy (Part 2): Multicenter Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Apr 30;6(4):e104. doi: 10.2196/mhealth.9438. PMID 29712622
- [Derived] Hsu HT, Yu CN, Sun WN, Liang TY, Weng SF, Yu E, Hsu YF. Feasibility and Acceptability of a Mobile App Intervention to Promote Self-Efficacy and Resilience Among Breast Cancer Patients Undergoing Chemotherapy: A Pilot Randomized Controlled Trial. Psychooncology. 2025 Nov;34(11):e70331. doi: 10.1002/pon.70331. PMID 41217167